CLINICAL TRIAL: NCT01929031
Title: A Single-centre, Double-blind, Randomised, Two-stage, Parallel-group Study to Assess the Efficacy and Safety of the Fixed Dose Combination of Ibuprofen 400 mg and Caffeine 100 mg Versus Ibuprofen 400 mg, Caffeine 100 mg and Placebo in Patients With Postoperative Dental Pain
Brief Title: Efficacy and Safety of Ibuprofen and Caffeine in Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1335.1
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Results first posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-09

CONDITIONS: Pain, Postoperative; Tooth Diseases
MeSH Terms: conditions — Pain, Postoperative; Tooth Diseases | interventions — Ibuprofen; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Caffeine-Ibuprofen (Other): Study Stage 1: One Caffeine 100 mg tablet after dental surgery; Arm Type: Active Comparator - Study Stage 2: Subsequent to Stage 1, every 6-8 hours one ibuprofen 400 mg tablet, while awake, over 5 days; Arm Type: Active Comparator
  Interventions: Drug: ibuprofen; Drug: caffeine
- Placebo-Ibuprofen/Caffeine (Other): Study Stage 1: One Placebo tablet after dental surgery Arm Type: Placebo Comparator - Study Stage 2: Subsequent to Stage 1, every 6-8 hours one Ibuprofen 400 mg/Caffeine tablet, while awake, over 5 days; Arm Type: Experimental
  Interventions: Drug: ibuprofen + caffeine; Drug: placebo
- Ibuprofen/Caffeine-Ibuprofen/Caffeine (Other): Study Stage 1: One Ibuprofen 400 mg/Caffeine 100 mg tablet after dental surgery: Arm Type Experimental - Study Stage 2: Subsequent to Stage 1, every 6-8 hours one Ibuprofen 400 mg/Caffeine 100 mg tablet, while awake, over 5 days; Arm Type Experimental
  Interventions: Drug: ibuprofen + caffeine
- Ibuprofen-Ibuprofen (Other): Study Stage 1: One Ibuprofen 400 mg tablet after dental surgery; Arm Type Active Comparator - Study Stage 2: Subsequent to stage 1, every 6-8 hours one Ibuprofen 400 mg tablet, while awake, over 5 days; Arm type; Active Comparator
  Interventions: Drug: ibuprofen
- Caffeine-Ibuprofen/Caffeine (Other): Study Stage 1: One Caffeine 100 mg tablet after dental surgery. Arm Type; Active Comparator - Study Stage 2: Subsequent to Stage 1, every 6-8 hours one Ibuprofen 400mg/Caffeine 100 mg tablet, while awake, over 5 days; Arm Type: Experimental
  Interventions: Drug: caffeine; Drug: ibuprofen + caffeine
- Placebo-Ibuprofen (Other): Study Stage 1: One Placebo tablet after dental surgery Arm Type: Placebo Comparator - Study Stage 2: Subsequent to Stage 1, every 6-8 hours one Ibuprofen 400 mg tablet, while awake over 5 days; Arm Type: Active Comparator
  Interventions: Drug: placebo; Drug: ibuprofen

INTERVENTIONS:
Drug: ibuprofen + caffeine — FDC tablet
  Arms: Placebo-Ibuprofen/Caffeine
Drug: ibuprofen — tablet.
  Arms: Ibuprofen-Ibuprofen
Drug: ibuprofen — tablet
  Arms: Caffeine-Ibuprofen
Drug: caffeine — tablet
  Arms: Caffeine-Ibuprofen/Caffeine
Drug: ibuprofen + caffeine — Fixed Dose Combination (FDC) tablet
  Arms: Ibuprofen/Caffeine-Ibuprofen/Caffeine
Drug: placebo — tablet
  Arms: Placebo-Ibuprofen
Drug: placebo — tablet
  Arms: Placebo-Ibuprofen/Caffeine
Drug: caffeine — tablet
  Arms: Caffeine-Ibuprofen
Drug: ibuprofen — tablet
  Arms: Placebo-Ibuprofen
Drug: ibuprofen + caffeine — FDC tablet
  Arms: Caffeine-Ibuprofen/Caffeine

SUMMARY:
The primary objective of this study is to compare the efficacy of a combination product containing ibuprofen 400 mg and caffeine 100 mg versus either ingredient alone as well as placebo for the treatment of post-surgical dental pain over an eight-hour period followed by a single dose of study medication (study stage 1). A secondary objective is to evaluate efficacy of multiple doses of the combination in comparison to ibuprofen alone over a 5-day post-surgical period (study stage 2).

ELIGIBILITY:
Inclusion criteria:

* Males and females 18 to 55 years of age;
* Outpatients scheduled to undergo surgical extraction of 3-4 impacted third molar(s), with a minimum of two mandibular extractions. The two mandibular third molars may be partial bony impactions or full bony impactions (as long as the trauma rating is not severe and the surgeons do not feel the subject will have extreme post-surgical pain) OR there may be a combination of one full bony impaction with the second mandibular being a soft tissue impaction or partial bony impaction. Maxillary third molars (or supernumerary teeth) of any type can be extracted;
* Use of only the following preoperative medication(s)/ anesthetic(s): topical benzocaine, short-acting local anesthetic (mepivacaine or lidocaine) with or without vasoconstrictor and/or nitrous oxide;
* Reliable, cooperative, and of adequate intelligence to record the requested information on the analgesic questionnaire form;
* Examined by the attending oral surgeon or physician and medically cleared to participate in the study;
* Scheduled to undergo a qualifying surgical procedure;
* In good general health, with a BMI of 30 or less, and have no contraindications to any of the study medications or anesthetic drugs;
* Subjects have at least a categorical pain score of moderate and a numerical rating scale (NRS) score of 5 or greater within 4.5 hours from the time of the last suture.

Exclusion criteria:

* Presence of a serious medical condition (e.g., poorly controlled hypertension, poorly controlled diabetes, significantly impaired cardiac, renal or hepatic function, hyper- or hypothyroidism);
* Use of a prescription or non-prescription drug with which the administration of ibuprofen or any other non steroidal anti inflammatory or caffeine is contraindicated;
* Acute local infection at the time of surgery that could confound the post-surgical evaluation;
* Females who are pregnant, lactating, of child-bearing potential, or post-menopausal for less than 2 years and not using a medically approved method of contraception (i.e., oral, transdermal, intravaginal or implanted contraceptives, intrauterine device, diaphragm, condom, abstinence, or surgical sterility), or females who test positive on a urine-based pregnancy test;
* Presence or history (within 2 years of enrollment) of bleeding disorder(s) or peptic ulcer disease;
* History of alcoholism or substance abuse within the last year, or is currently abusing alcohol or other mood-altering drugs (e.g., cannabis). Subjects who are taking central nervous system or other psychotropic drugs (including St. Johns Wort, or any other nutritional supplement known to have psychotropic effects) may be enrolled if they have been on stable doses of medication for at least 2 months, will maintain this dose throughout the study, and their condition is judged by the Principal Investigator to be well-controlled;
* Habituation to analgesic drugs or caffeine (i.e., routine use of oral analgesics 5 or more times per week or ingestion of 4 or more caffeine-containing drinks daily); use of "high energy" drinks more than once per week;
* Use of any type of systemic corticosteroid within the past 30 days or a history of current or previous use of anabolic steroids;
* History of allergic reaction (e.g., asthma, rhinitis, swelling, shock, or hives) to acetaminophen, ibuprofen, naproxen, aspirin, celecoxib, or any other non steroidal anti inflammatory or caffeine;
* Prior use of any type of analgesic or non steroidal anti inflammatory within 5 half-lives of that drug before surgery, except for pre-anesthetic medication and anesthesia for the procedure;
* Ingestion of any caffeine-containing beverages, chocolate, or alcohol 6 hours or less before surgery;
* Has impaired liver function, e.g., serum Alanine transaminase, aspartate aminotransferase, alkaline phosphatase, or Gamma-glutamyltransferase greater than 2.5 times the upper limit of normal, or blood urea nitrogen, creatinine, or bilirubin greater than 1.5 times the upper limit of normal without a known benign explanation;
* Has known history of a positive HIV antibody test or known HIV infection;
* Has a known history of Hepatitis B or C;
* Has a clinically significant abnormal electrocardiogram (ECG) at screening as determined by the Investigator:
* Has taken an investigational product within the past 30 days;
* Has previously been entered into this study;
* The subject is a member of the study site staff either directly involved with the study, an employee of the Sponsor, or a relative of study site personnel directly involved with the study or Sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 562 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1335.1.202 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Forderreuther S, Lampert A, Hitier S, Lange R, Weiser T. The Impact of Baseline Pain Intensity on the Analgesic Efficacy of Ibuprofen/Caffeine in Patients with Acute Postoperative Dental Pain: Post Hoc Subgroup Analysis of a Randomised Controlled Trial. Adv Ther. 2020 Jun;37(6):2976-2987. doi: 10.1007/s12325-020-01297-y. Epub 2020 Apr 24. PMID 32333328
- [Derived] Weiser T, Richter E, Hegewisch A, Muse DD, Lange R. Efficacy and safety of a fixed-dose combination of ibuprofen and caffeine in the management of moderate to severe dental pain after third molar extraction. Eur J Pain. 2018 Jan;22(1):28-38. doi: 10.1002/ejp.1068. Epub 2017 Aug 14. PMID 28805281

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibuprofen/Caffeine - Ibuprofen/Caffeine: Study stage 1: One Ibuprofen 400mg/Caffeine 100mg tablet after dental surgery; Study stage 2: Subsequent to stage 1, every 6-8 hours one Ibuprofen400mg/Caffeine 100mg tablet, while awake, over 5 days
- Ibuprofen - Ibuprofen: Study stage 1: One Ibuprofen 400mg tablet after dental surgery; Study stage 2: Subsequent to stage 1, every 6-8 hours one Ibuprofen 400mg tablet, while awake, over 5 days
- Caffeine - Ibuprofen/Caffeine: Study stage 1: One Caffeine 100mg tablet after dental surgery; Study stage 2: Subsequent to stage 1, every 6-8 hours one Ibuprofen 400mg/Caffeine 100mg tablet, while awake, over 5 days
- Caffeine - Ibuprofen: Study stage 1: One Caffeine 100mg tablet after dental surgery; Study stage 2: Subsequent to stage 1, every 6-8 hours one Ibuprofen 400mg tablet, while awake, over 5 days
- Placebo - Ibuprofen/Caffeine: Study stage 1: One Placebo tablet after dental surgery; Study stage 2: Subsequent to stage 1, every 6-8 hours one Ibuprofen 400mg/Caffeine 100mg tablet, while awake, over 5 days
- Placebo - Ibuprofen: Study stage 1: One Placebo tablet after dental surgery; Study stage 2: Subsequent to stage 1, every 6-8 hours one Ibuprofen 400mg tablet, while awake, over 5 days
Period: Overall Study
Arm/Group | Ibuprofen/Caffeine - Ibuprofen/Caffeine | Ibuprofen - Ibuprofen | Caffeine - Ibuprofen/Caffeine | Caffeine - Ibuprofen | Placebo - Ibuprofen/Caffeine | Placebo - Ibuprofen
Started | 213 | 209 | 35 | 35 | 34 | 36
Completed | 209 | 207 | 34 | 35 | 33 | 35
Not Completed | 4 | 2 | 1 | 0 | 1 | 1
Not completed — Adverse Event | 3 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Reason other than specified above | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated patients
Groups:
- Placebo Stage 1: One Placebo tablet after dental surgery
- Caffeine Stage 1: One Caffeine 100mg tablet after dental surgery
- Ibuprofen Stage 1: One Ibuprofen 400mg tablet after dental surgery
- Ibuprofen/Caffeine Stage 1: One Ibuprofen 400mg/Caffeine 100mg tablet after dental surgery
- Total: Total of all reporting groups
Arm/Group | Placebo Stage 1 | Caffeine Stage 1 | Ibuprofen Stage 1 | Ibuprofen/Caffeine Stage 1 | Total
Number analyzed (Participants) | 70 | 70 | 209 | 213 | 562
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.3 (1.77) | 19.2 (1.72) | 19.6 (1.96) | 19.5 (2.06) | 19.5 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 39 | 142 | 131 | 358
  Male | 24 | 31 | 67 | 82 | 204
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 209 | 213 | 562

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Relief (PAR) and Pain Intensity Difference (PID) From 0 to 8 Hours (SPRID0-8h)
Description: SPRID0-8h: Time-weighted sum of PAR and PID from 0 to 8 hours, score range: -40 (worst) to 112 (best). PI was assessed on a 0-10 numerical pain rating scale (NPRS), where 0=no pain and 10=worst possible pain, pre-dose and at 0.25,0.5,0.75,1,1.5,2,3,4,5, 6,7 and 8 hours; PAR was assessed on a 5-point verbal rating scale (VRS) (0=none to 4=complete) at the same post-dose time points. Time-weights were equal to the elapsed time (hour) between the time point of interest and the preceding time point. All PAR and pain intensity (PI) assessments completed after the patient had taken rescue medication or the second dose of study medication, whichever was first, until hour 8 were considered missing. Last observation carried forward (LOCF) was used with the last completed PI/PAR assessments prior to first rescue/second study medication, whichever was first, to impute missing values up to 8 hours.
Time Frame: 0 to 8 hours
Population: Randomized patients who used at least one dose of study medication and provided any post-treatment data for the primary efficacy endpoint (FAS)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: One Placebo tablet after dental surgery
- Caffeine: One Caffeine 100mg tablet after dental surgery
- Ibuprofen: One Ibuprofen 400mg tablet after dental surgery
- Ibuprofen/Caffeine: One Ibuprofen 400mg/Caffeine 100mg tablet after dental surgery
Arm/Group | Placebo | Caffeine | Ibuprofen | Ibuprofen/Caffeine
Number analyzed (Participants) | 70 | 70 | 209 | 213
units on a scale | 10.554 (3.527) | 15.824 (3.525) | 40.165 (2.047) | 52.291 (2.027)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen/Caffeine; Test type: Superiority or Other; p < 0.0001, ANCOVA; The statistical model included baseline PI (VRS), and treatment; Mean Difference (Final Values) = 41.738, 95% CI 2-sided [33.767 to 49.708], Standard Error of Mean 4.058 — Ibuprofen/Caffeine vs. Placebo
Statistical Analysis 2: Comparison: Caffeine vs Ibuprofen/Caffeine; Test type: Superiority or Other; p < 0.0001, ANCOVA; The statistical model included baseline PI (VRS), and treatment; Mean Difference (Final Values) = 36.467, 95% CI 2-sided [28.497 to 44.437], Standard Error of Mean 4.058 — Ibuprofen/Caffeine vs. Caffeine
Statistical Analysis 3: Comparison: Ibuprofen vs Ibuprofen/Caffeine; Test type: Superiority or Other; p < 0.0001, ANCOVA; The statistical model included baseline PI (VRS), and treatment; Mean Difference (Final Values) = 12.126, 95% CI 2-sided [6.493 to 17.759], Standard Error of Mean 2.868 — Ibuprofen/Caffeine vs. Ibuprofen

2. Secondary Outcome: Time-weighted Sum of Pain Relief (PAR) and Pain Intensity Difference (PID) From 0 to 2 Hours (SPRID0-2h)
Description: SPRID0-2h: Time-weighted sum of PAR and PID from 0 to 2 hours, score range: -10 (worst) to 28 (best). PI was assessed on a 0-10 numerical pain rating scale (NPRS), where 0=no pain and 10=worst possible pain, pre-dose and at 0.25,0.5,0.75,1,1.5 and 2 hours; PAR was assessed on a 5-point verbal rating scale (VRS) (0=none to 4=complete) at the same post-dose time points. Time-weights were equal to the elapsed time (hour) between the time point of interest and the preceding time point. All PAR and pain intensity (PI) assessments completed after the patient had taken rescue medication or the second dose of study medication, whichever was first, until hour 2 was considered missing. Last observation carried forward (LOCF) was used with the last completed PI/PAR assessments prior to first rescue/second study medication, whichever was first, to impute missing values up to 2 hours.
Time Frame: 0 to 2 hours
Population: Patients who used at least one dose of study medication and provided any post-treatment data for the primary efficacy endpoint (FAS)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Caffeine | Ibuprofen | Ibuprofen/Caffeine
Number analyzed (Participants) | 70 | 70 | 209 | 213
units on a scale | 2.059 (0.703) | 2.612 (0.702) | 6.990 (0.408) | 10.584 (0.404)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen/Caffeine; Test type: Superiority or Other; p < 0.0001, ANCOVA; The statistical model included baseline PI (VRS), and treatment; Mean Difference (Final Values) = 8.525, 95% CI 2-sided [6.937 to 10.113], Standard Error of Mean 0.808 — Ibuprofen/Caffeine vs. Placebo
Statistical Analysis 2: Comparison: Caffeine vs Ibuprofen/Caffeine; Test type: Superiority or Other; p < 0.0001, ANCOVA; The statistical model included baseline PI (VRS), and treatment; Mean Difference (Final Values) = 7.972, 95% CI 2-sided [6.384 to 9.559], Standard Error of Mean 0.808 — Ibuprofen/Caffeine vs. Caffeine
Statistical Analysis 3: Comparison: Ibuprofen vs Ibuprofen/Caffeine; Test type: Superiority or Other; p < 0.0001, ANCOVA; The statistical model included baseline PI (VRS), and treatment; Mean Difference (Final Values) = 3.594, 95% CI 2-sided [2.472 to 4.716], Standard Error of Mean 0.571 — Ibuprofen/Caffeine vs. Ibuprofen

3. Secondary Outcome: Duration of Pain Relief
Description: Duration of pain relief was defined as the time between the administration of first dose of trial medication and first dose of rescue medication or second dose of trial medication, whichever was first. Duration of pain relief was censored at 8 hours.
Time Frame: 8 hours
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Caffeine | Ibuprofen | Ibuprofen/Caffeine
Number analyzed (Participants) | 70 | 70 | 209 | 213
hours | 1.63 [1.60 to 2.07] | 2.08 [1.67 to 3.83] | 7.11 [6.43 to 7.77] | 7.33 [7.05 to 7.77]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen/Caffeine; Ibuprofen/Caffeine vs. Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank; Log rank test stratified for baseline pain intensity as measured on the 4-point VRS
Statistical Analysis 2: Comparison: Caffeine vs Ibuprofen/Caffeine; Ibuprofen/Caffeine vs. Caffeine; Test type: Superiority or Other; p < 0.0001, Log Rank; Log rank test stratified for baseline pain intensity as measured on the 4-point VRS
Statistical Analysis 3: Comparison: Ibuprofen vs Ibuprofen/Caffeine; Ibuprofen/Caffeine vs. Ibuprofen; Test type: Superiority or Other; p = 0.2389, Log Rank; Log rank test stratified for baseline pain intensity as measured on the 4-point VRS

4. Secondary Outcome: Time to Meaningful Pain Relief
Description: Time to meaningful pain relief was captured by a stopwatch, which was started by the study staff immediately after the administration of the first dose of trial medication and which was to be stopped by the patient as soon as he/she felt meaningful pain relief. Time to meaningful pain relief was censored at 8 hours.
Time Frame: 8 hours
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Caffeine | Ibuprofen | Ibuprofen/Caffeine
Number analyzed (Participants) | 70 | 70 | 209 | 213
hours | NA [NA to NA] — because more than half of the patients were without meaningful pain relief within 8 h | NA [NA to NA] — because more than half of the patients were without meaningful pain relief within 8 h | 1.78 [1.48 to 2.02] | 1.13 [0.93 to 1.35]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen/Caffeine; Ibuprofen/Caffeine vs. Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank; Log rank test stratified for baseline pain intensity as measured on the 4-point VRS
Statistical Analysis 2: Comparison: Caffeine vs Ibuprofen/Caffeine; Ibuprofen/Caffeine vs. Caffeine; Test type: Superiority or Other; p < 0.0001, Log Rank; Log rank test stratified for baseline pain intensity as measured on the 4-point VRS
Statistical Analysis 3: Comparison: Ibuprofen vs Ibuprofen/Caffeine; Ibuprofen/Caffeine vs. Ibuprofen; Test type: Superiority or Other; p = 0.0001, Log Rank; Log rank test stratified for baseline pain intensity as measured on the 4-point VRS

ADVERSE EVENTS:
Time Frame: First dose of study drug date/time until drug discontinuation date + 24 hours (inclusive)
Description: Patients at risk and reported adverse events were allocated to the actual treatment patients were exposed to, regardless of the study stage.
Groups:
- Placebo: Placebo tablet
- Caffeine: Caffeine 100mg tablet
- Ibuprofen: Ibuprofen 400mg tablet
- Ibuprofen/Caffeine: Ibuprofen 400mg / Caffeine 100mg tablet
Arm/Group | Placebo | Caffeine | Ibuprofen | Ibuprofen/Caffeine
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70 | 1/279 | 0/282
Other Adverse Events (participants affected / at risk) | 3/70 | 1/70 | 9/279 | 23/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=70) | Caffeine (N=70) | Ibuprofen (N=279) | Ibuprofen/Caffeine (N=282)
Oral infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=70) | Caffeine (N=70) | Ibuprofen (N=279) | Ibuprofen/Caffeine (N=282)
Nausea (Gastrointestinal disorders) | 3 | 1 | 9 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.